CLINICAL TRIAL: NCT00977561
Title: A Phase 2, Randomized, Open Label Study Of Figitumumab (CP-751,871) Plus Cisplatin (Or Carboplatin) And Etoposide, Versus Cisplatin (Or Carboplatin) And Etoposide Alone, As First Line Treatment In Patients With Extensive Stage Disease Small Cell Lung Cancer
Brief Title: A Study Of Cisplatin (Or Carboplatin) And Etoposide With Or Without Figitumumab (CP-751,871) In Patients With Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021032
Record Dates: First submitted 2009-09-10; First posted 2009-09-15 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-01

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Small Cell Lung Cancer; Extensive stage disease; SCLC; IGF-1R inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — figitumumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Figitumumab (CP-751,871) Plus Chemotherapy [Cisplatin (Or Carboplatin) And Etoposide] All drugs to be administered on a 21 day cycle
  Interventions: Drug: figitumumab; Drug: Cisplatin (Or Carboplatin); Drug: Etoposide
- Arm B (Active Comparator): Chemotherapy [Cisplatin (Or Carboplatin) And Etoposide] All drugs to be administered on a 21 day cycle
  Interventions: Drug: Cisplatin (Or Carboplatin); Drug: Etoposide

INTERVENTIONS:
Drug: figitumumab — Figitumumab (20 mg/kg)
  Arms: Arm A
Drug: Cisplatin (Or Carboplatin) — Cisplatin (75 mg/m2 IV on Day 1) or Carboplatin AUC 5
  Arms: Arm A
Drug: Etoposide — Etoposide (100 mg/m2 IV on Days 1, 2 and 3)
  Arms: Arm A
Drug: Cisplatin (Or Carboplatin) — Cisplatin (75 mg/m2 IV on Day 1) or Carboplatin AUC 5
  Arms: Arm B
Drug: Etoposide — Etoposide (100 mg/m2 IV on Days 1, 2 and 3)
  Arms: Arm B

SUMMARY:
This study will summarize the safety of patients receiving figitumumab combined with etoposide and cisplatin (or carboplatin) vs. patients receiving etoposide and cisplatin (or carboplatin) alone as first line treatment for extensive stage disease Small Cell Lung Cancer.

DETAILED DESCRIPTION:
The study prematurely discontinued on January 26, 2011 due to slow enrollment. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of extensive stage disease Small Cell Lung Cancer (SCLC), with tumor biopsy sample required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. Total IGF-1 > or = 120 ng/ml

Exclusion Criteria:

* Any prior systemic therapy for Small Cell Lung Cancer (SCLC)
* HbA1c > or = 5.7%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (31):
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Lenoir, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, Mount Airy, North Carolina
  - Pfizer Investigational Site, North Wilkesboro, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Beaverton, Oregon
  - Pfizer Investigational Site, Gresham, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Tualatin, Oregon
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Christiansburg, Virginia
  - Pfizer Investigational Site, Low Moor, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Salem, Virginia
  - Pfizer Investigational Site, Wytheville, Virginia
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Gig Harbor, Washington
  - Pfizer Investigational Site, Kennewick, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Canada (4):
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Hungary (5):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Farkasgyepű
  - Pfizer Investigational Site, Törökbálint
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021032&StudyName=A%20Study%20Of%20Cisplatin%20%28Or%20Carboplatin%29%20And%20Etoposide%20With%20Or%20Without%20Figitumumab%20%28CP-751%2C871%29%20In%20Patients%20With%20Extensive-Stage%20Smal

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab + Cisplatin or Carboplatin + Etoposide: Figitumumab 20 milligram/kilogram (mg/kg) administered intravenously (IV) over 1 hour on Day 2 of Cycle 1 and on Day 1 of subsequent cycles (up to 17 cycles in the absence of further disease progression or intolerable toxicity). Cisplatin 75 milligram/square meter (mg/m^2) IV over 1 hour or carboplatin at a dose to attain the target area under the concentration-time curve (AUC) of 5 milligram/milliliter*minute (mg/mL*min) IV over 15-60 minutes on Day 1 (up to 6 cycles) followed by etoposide 100 mg/m^2 IV over 1 hour on Days 1, 2 and 3 of each cycle (up to 6 cycles or until progression or intolerable toxicity). Each cycle was 21 days cycle.
- Cisplatin or Carboplatin + Etoposide: Cisplatin 75 mg/m^2 IV over 1 hour or carboplatin at a dose to attain the target AUC of 5 mg/mL*min IV over 15-60 minutes on Day 1 (up to 6 cycles) followed by etoposide 100 mg/m^2 IV over 1 hour on Days 1, 2 and 3 of each cycle (up to 6 cycles or until progression or intolerable toxicity). Each cycle was 21 days cycle.
Period: Overall Study
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Started | 5 | 4
Completed | 0 | 0
Not Completed | 5 | 4
Not completed — Death | 3 | 2
Not completed — Study terminated | 0 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Figitumumab + Cisplatin or Carboplatin + Etoposide: Figitumumab 20 mg/kg administered IV over 1 hour on Day 2 of Cycle 1 and on Day 1 of subsequent cycles (up to 17 cycles in the absence of further disease progression or intolerable toxicity). Cisplatin 75 mg/m^2 IV over 1 hour or carboplatin at a dose to attain the target AUC of 5 mg/mL*min IV over 15-60 minutes on Day 1 (up to 6 cycles) followed by etoposide 100 mg/m^2 IV over 1 hour on Day 1, 2 and 3 of each cycle (up to 6 cycles or until progression or intolerable toxicity). Each cycle was 21 days cycle.
- Total: Total of all reporting groups
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide | Total
Number analyzed (Participants) | 5 | 4 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (4.4) | 53.8 (11.0) | 57.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Median time from the first dose of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. PFS time (days) = [event (progression or death) date or censor date - date of randomization + 1].
Time Frame: Baseline, every 2nd cycle (between Day 15-21, 1 cycle = 21 days) starting with Cycle 2 until disease progression, at the end of treatment visit (if more than 28 days have passed since last evaluation); and every 6 weeks until disease progression
Population: No analysis of progression-free survival was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Groups:
- Figitumumab + Cisplatin or Carboplatin + Etoposide: Figitumumab 20 mg/kg administered IV over 1 hour on Day 2 of Cycle 1 and on Day 1 of subsequent cycles (up to 17 cycles in the absence of further disease progression or intolerable toxicity). Cisplatin 75 mg/m^2 IV over 1 hour or carboplatin at a dose to attain the target AUC of 5 mg/mL*min IV over 15-60 minutes on Day 1 (up to 6 cycles) followed by etoposide 100 mg/m^2 IV over 1 hour on Days 1, 2 and 3 of each cycle (up to 6 cycles or until progression or intolerable toxicity). Each cycle was 21 days cycle.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as ≥30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST.
Time Frame: as for outcome 1
Population: No analysis of objective response was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was the duration from enrollment to death due to any cause. For participants who are alive, overall survival was censored at the last contact. Survival time (days) = [death date (last known alive date) - date of randomization +1].
Time Frame: Every 3 months until death or 12 months from the date the last participant was randomized
Population: No analysis of overall survival was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs are any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study treatment. The event does not need to be causally related to the study treatment. SAEs include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly or birth defect in the offspring of a study subject.
Time Frame: Baseline up to follow-up (90 days post dose)
Population: All randomized participants who received at least one dose of any agent of the combination were included in the safety analysis.
Measure: Number; unit: participants
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 5 | 4
participants
  Adverse Events | 5 | 4
  Serious Adverse Events | 4 | 2

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Figitumumab
Time Frame: Cycle 1, Day 2; Day 1 of Cycles 2, 4, 5, 6, 10 and 15; Day 28 and Day 90 post last figitumumab dose
Population: No analysis of Cmax for figitumumab was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Groups:
- Figitumumab+ Cisplatin (or Carboplatin) + Etoposide: Figitumumab 20 mg/kg administered IV over 1 hour on Day 2 of Cycle 1 and on Day 1 of subsequent cycles (up to 17 cycles in the absence of further disease progression or intolerable toxicity). Cisplatin 75 mg/m^2 IV over 1 hour or carboplatin at a dose to attain the target AUC of 5 mg/mL*min IV over 15-60 minutes on Day 1 (up to 6 cycles) followed by etoposide 100 mg/m^2 IV over 1 hour on Days 1, 2 and 3 of each cycle (up to 6 cycles or until progression or intolerable toxicity). Each cycle was 21 days cycle.
Arm/Group | Figitumumab+ Cisplatin (or Carboplatin) + Etoposide
Number analyzed (Participants) | 0

6. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of Figitumumab
Time Frame: Cycle 1, Day 2; Day 1 of Cycles 2, 4, 5, 6, 10 and 15; Day 28 and Day 90 post last figitumumab dose
Population: No analysis of Cmin for figitumumab was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Etoposide
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Cycles 1 and 2, Day 1 and Day 2 (within 3 hours prior to Day 1 etoposide infusion; 1, 1.5, 2, 3, 6, and 24 hours post Day 1 etoposide infusion); Cycles 4 and 5, Day 2: 24 hours post Day 1 etoposide infusion
Population: No analysis of pharmacokinetics (PK) parameters for etoposide was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Etoposide
Time Frame: as for outcome 7
Population: No analysis of PK parameters for etoposide was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants Reporting Positive Anti-Drug Antibodies (ADA) Response for Figitumumab
Description: Percentage of participants with positive total or neutralizing anti-drug antibody (ADA) for figitumumab
Time Frame: Day 2 of Cycle 1 (or Day 1 of the initial cycle starting single agent figitumumab); Day 1 of Cycles 2 and 4; Day 28 and Day 90 post last figitumumab dose
Population: No analysis of ADA response was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Groups:
- Figitumumab + Cisplatin or Carboplatin + Etoposide: Participants who received figitumumab, whether figitumumab (20 mg/kg, IV over 1 hour on Day 2 of Cycle 1 and on Day 1 of subsequent cycles) was given in combination with cisplatin (75 mg/m^2 IV over 1 hour on Day 1 of each cycle) or carboplatin (AUC of 5 mg/mL*min IV over 15-60 minutes on Day 1 of each cycle) followed by etoposide (100 mg/m^2 IV over 1 hour on Days 1, 2 and 3 of each cycle) from the beginning or figitumumab was given as a single agent after documented disease progression with cisplatin (or carboplatin) and etoposide. When given as a single agent, figitumumab was administered as IV infusion on Days 1 and 2 of the initial cycle and on Day 1 of subsequent cycles, up to 17 cycles in the absence of further disease progression or intolerable toxicity. Each cycle was 21 days cycle.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0

10. Secondary Outcome: Cancer Dyspnea Scale (CDS) Score
Description: The Cancer Dyspnea Scale consists of 12 questions that assess 3 domains of dyspnea (sense of effort, anxiety and discomfort) related to lung cancer. The questions are answered on 5-point Likert scale ranging from 1 to 5 (1 "Not at All" to 5 "Very Much").
Time Frame: Day 1 of every cycle (up to 17 cycles), at the end of treatment visit (28 days post last dose); then every 6 weeks until disease progression
Population: No analysis for cancer dyspnea scale score was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Numeric Rating Scale (NRS) Score
Description: The Numeric Rating Scale (NRS) is a 1-item self-reported questionnaire designed to assess "worst pain" severity. Overall scores range from 0 to 10, with low scores representing a lower level of pain.
Time Frame: as for outcome 10
Population: No analysis for NRS score was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Pre-treatment Levels of Tumor Biomarkers Involved in Insulin-Like Growth Factor 1 (IGF-I) Signaling Pathway
Time Frame: Baseline prior to dosing
Population: No analysis of tumor biomarkers was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Levels of Serum Circulating Insulin-like Growth Factor (IGF) Pathway Related Markers
Time Frame: Baseline (Cycle 1, Day 1 prior to dosing), Cycle 4 (Day 1), at the end of treatment visit (28 days post last figitumumab dose)
Population: No analysis for serum circulating IGF pathway related markers was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Total Circulating Tumor-Related Cells (CTCs) and Insulin-Like Growth Factor 1 Receptor (IGF-IR)-Expressing CTCs
Description: Pre-treatment and post-treatment counts of total and IGF-IR-positive CTCs
Time Frame: Baseline (Cycle 1, Day 1), Cycle 4 (Day 1) and at the end of treatment visit (28 days post last figitumumab dose)
Population: No analysis of total CTCs and IGF-IR-expressing CTCs was performed as the study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. As a result, the only endpoint analyzed for the study was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab + Cisplatin or Carboplatin + Etoposide | Cisplatin or Carboplatin + Etoposide
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Cisplatin or Carboplatin + Etoposide (N=5) | Cisplatin or Carboplatin + Etoposide (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab + Cisplatin or Carboplatin + Etoposide (N=5) | Cisplatin or Carboplatin + Etoposide (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 2 | 0
Feeling cold (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 2
Otitis media (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to low participants enrollment and the halting of the figitumumab development program. The only endpoint analyzed was safety and tolerability of figitumumab ± cisplatin (or carboplatin) and etoposide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.